CLINICAL TRIAL: NCT02061345
Title: A PET Imaging Study to Detect the Presence of Activated Microglia in the Brains of Prostate Cancer Patients Who Develop Mild Cognitive Impairment Following Androgen Deprivation Therapy
Brief Title: PET Imaging in MCI Following ADT for PCa
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 13HH0558
Record Dates: First submitted 2014-02-11; First posted 2014-02-12 (Estimated); Results first posted 2023-12-07 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-11

CONDITIONS: Prostate Cancer; Mild Cognitive Impairment
Keywords: Prostate cancer; Androgen Deprivation Therapy; Mild Cognitive Impairment
MeSH Terms: conditions — Prostatic Neoplasms; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples for determining TSPO (Ala147Thr) polymorphism, testosterone and estrogen hormone levels
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- MCI: Prostate cancer patients having mild cognitive impairment (MCI) attributable to ADT with LHRHa
- Control: Prostate cancer patients on ADT with LHRHa not having mild cognitive impairment

SUMMARY:
Mild cognitive impairment (MCI) with ageing is thought in part to be related to reduced serum sex hormones which is well-recognized, especially in females, but poorly understood. International studies assessing hormone replacement therapy (HRT) to prevent/reduce MCI are ongoing. MCI leads to morbidity, reduced quality of life and substantial healthcare costs. The commonest therapeutically induced reduction in sex hormone level in men is treatment of prostate cancer (PCa). PCa is androgen dependent and androgen deprivation therapy (ADT) suppressing testosterone to castrate levels is key therapy for advanced disease. About one million men worldwide have received ADT for PCa, mostly using luteinising hormone releasing hormone agonists (LHRHa) although oral oestrogens were used in the past; eventually perhaps 4% of Caucasians may be castrated. MCI as a side effect of castration in men remains poorly researched. This study aims to demonstrate that pathological changes occur in the brains of a significant proportion of prostate cancer patients subjected to ADT that correlate with MCI symptoms. Highlighting the pathological changes of MCI should improve understanding and interventions for slowing/preventing MCI in PCa survivors. Brain scans employing positron emission tomography (PET) imaging technique will be used to detect the presence of pathological changes in the brain that relate to ADT induced MCI. MCI will be assessed by neuropsychological assessments (standard paper-based questionnaires and online) and its neural basis will be investigated using magnetic resonance imaging (MRI).

DETAILED DESCRIPTION:
In males, MCI with aging is thought in part to be related to reduction in serum androgen level and international studies are on-going to prevent age-related cognitive decline using androgen replacement therapy. Reduction in cognitive function often leads to morbidity and reduction in quality of life. The commonest therapeutically induced reduction in sex hormone level in men is in the treatment of prostate cancer. As prostate cancer is androgen dependent for growth, androgen-deprivation therapy (ADT) to suppress serum testosterone level to castration levels (< 1.7mM) is the key therapeutic intervention for advanced disease. Up to 1 million men worldwide are estimated to have been prescribed ADT for prostate cancer, mostly using luteinising hormone releasing hormone agonists (LHRHa). ADT is now also used to treat some early prostate cancer and as early asymptomatic prostate cancer is increasingly being diagnosed and treated following screening with serum prostate-specific antigen (PSA) measurement, estimates suggest that eventually up to 4% of all Caucasians will be castrated, some of them remaining on ADT for as long as 10 years or more. ADT is associated with considerable adverse effects, including MCI. Up to 69% of men showed MCI after six to nine months of ADT, with a decline in at least one cognitive area, most commonly visuospatial ability and executive function. Little work has been done to quantify MCI due to ADT, understand the mechanism, predict which patients will be affected and determine ways of reducing this side effect.

Establishing the presence of pathophysiology in ADT induced MCI first is important due to the lack of understanding of the underlying mechanism. A plausible scientific approach in this regard appears to be the use of the brain's immunological response to pathology using a PET imaging ligand for activated microglia. Brain microglia have been demonstrated to be highly responsive to brain injury and are rapidly activated in an attempt to envelope/ contain the focal pathology. When activated, brain microglia have been shown to express the translocator protein (TSPO). The 18 kilo-Dalton (KDa) translocator protein (TSPO) formerly known as the peripheral benzodiazepine receptor (PBR) is widely expressed in the body but is particularly enriched up to 20 to 50 fold in steroid synthesising tissues. High TSPO expression has also been reported in immune cells such as macrophages and monocytes and TSPO is a well-characterised marker of neuroinflammation. PET imaging ligands have been developed for TSPO and used successfully for researching a range of brain disorders. While such imaging does not provide mechanistic information of the underlying pathology, except for the exasperation of frank neuro-inflammation, it does offer a generic sensitive bio-marker for demonstrating the presence of an on-going active pathology

ELIGIBILITY:
Inclusion Criteria:

1. Prostate cancer patients between the ages 50 to 80 years on ADT with LHRHa for for 3 months up to a year.
2. Able to give written informed consent.
3. Able to lie still for up to 90 minutes for a PET scan.
4. Not claustrophobic and so able to undergo an MRI scan.

Exclusion Criteria:

1. Patients with a known history of organic brain disorders and associated dementia, delirium and other specific neuropsychiatric conditions, including stroke and head injury.
2. Patients who are clinically assessed as having MCI prior to starting ADT.
3. Patients with a medical prognosis of less than 3 months.
4. Patients who are claustrophobic.
5. Patients who have any metal implanted in their body e.g. heart pacemaker, cochlear implant or any other electronic device.

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 12 prostate cancer patients on ADT with LHRHa will be recruited for the imaging part of the study; six patients having significant cognitive impairment attributable to LHRHa and six patients without cognitive impairment.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2014-04; Primary Completion 2016-12 (Actual); Study Completion 2022-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul D Abel, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

REFERENCES:
- [Result] Saleem A, Shah SIA, Mangar SA, Coello C, Wall MB, Rizzo G, Jones T, Price PM. Cognitive Dysfunction in Patients Treated with Androgen Deprivation Therapy: A Multimodality Functional Imaging Study to Evaluate Neuroinflammation. Prostate Cancer. 2023 Oct 18;2023:6641707. doi: 10.1155/2023/6641707. eCollection 2023. PMID 37885823

RESULTS

PARTICIPANT FLOW:
Groups:
- Mild Cognitive Impairment MCI: Prostate cancer patients having mild cognitive impairment (MCI) attributable to ADT with LHRHa
Period: Overall Study
Arm/Group | Mild Cognitive Impairment MCI | Control
Started | 6 | 5
Completed | 6 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mild Cognitive Impairment MCI | Control | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 5 | 4 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 6 | 5 | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: PET Biomarker Uptake
Description: The outcome measure is the increased uptake of 11-Carbon Peripheral Benzodiazepine Receptor-28 ([11C]PBR28) biomarker by activated microglia of patients demonstrating significant MCI with the primary endpoint of [11C]PBR28 uptake measured as a standardized uptake value (SUV)
Time Frame: Single time-point SUV in Hippocampus area on the day of the test
Measure: Mean (Standard Deviation); unit: Standard Uptake Measure SUV
Arm/Group | Mild Cognitive Impairment MCI | Control
Number analyzed (Participants) | 6 | 5
Standard Uptake Measure SUV | 0.95 (0.25) | 0.98 (0.18)

2. Secondary Outcome: PET Biomarker Volume of Distribution
Description: Secondary endpoint is the [11C]PBR28 total volume of distribution (VT)
Time Frame: Single time-point
Population: Data not collected
Arm/Group | Mild Cognitive Impairment MCI | Control
Number analyzed (Participants) | 0 | 0

3. Other Pre Specified Outcome: Cognitive Impairment
Description: Association of cognitive and neuropsychiatric impairments following ADT with structural and/or functional brain connectivity
Time Frame: Single time-point
Population: Data not collected
Arm/Group | Mild Cognitive Impairment MCI | Control
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: On day of imaging study
Arm/Group | Mild Cognitive Impairment MCI | Control
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/5
Other Adverse Events (participants affected / at risk) | 0/6 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2014-09-18): https://cdn.clinicaltrials.gov/large-docs/45/NCT02061345/Prot_000.pdf